CLINICAL TRIAL: NCT05520658
Title: Evaluation of the Efficacy of Intralesional Injection of Combined Digoxin and Furosemide Versus 5 - Fluorouracil in Treatment of Plantar Warts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Samah Ragab Ahmed, resident doctor at dermatology department at sohag teaching hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-07-01
Record Dates: First submitted 2022-08-15; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Plantar Wart
MeSH Terms: interventions — Furosemide; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): patients will receive intralesional combined digoxin and furosemide , one session every 2 weeks for maximum 6 sessions
  Interventions: Drug: combined digoxin and furosemide
- group B (Active Comparator): patients will receive intralesional 5 fluorouracil mixed with 1ml of 2% lignocaine and epinephrine one session every 2 weeks for maximum 6 sessions .
  Interventions: Drug: 5 fluorouracil

INTERVENTIONS:
Drug: combined digoxin and furosemide — one session every 2 weeks for maximum 6 sessions
  Arms: group A
Drug: 5 fluorouracil — 5 fluorouracil mixed with1ml of 2% lignocaine and epinephrine one session every 2 weeks for maximum 6 sessions .
  Arms: group B

SUMMARY:
Warts are common skin infections caused by human papillomavirus (HPV), which can cause a variety of skin presentations according to its type, site and the immune status .Nongenital warts may be presented as common, plane, plantar, filiform, or mucosal warts .Most people are affected by cutaneous warts, either plantar warts or common warts .prevalence of skin warts is between 3% and 13% and plantar warts are about 30% of skin warts in western world .Majority of cases occur in adolescent and young adults

ELIGIBILITY:
Inclusion Criteria:

* Age:>18 years .
* Sex: both males and females will be included.
* Confirmed diagnosis by clinical and dermoscopic examination of plantar warts will be made

Exclusion Criteria:

* Patients with history or evidenced hypersensitivity to any component used in this study.
* Pregnancy & lactating.
* Patients who receive immune suppressive therapy.
* Patients who receive any wart treatment during the last 2 months before enrollment in the study.
* Patients with systemic illness especially cardiac patients.
* Patients who refused participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
the change in size of plantar wart | 3 month
  measurement the change in size of plantar wart
the change in number of plantar warts | 3 month
  measurement the change in number of plantar warts

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abeck D, Tetsch L, Luftl M, Biedermann T. Extragenital cutaneous warts - clinical presentation, diagnosis and treatment. J Dtsch Dermatol Ges. 2019 Jun;17(6):613-634. doi: 10.1111/ddg.13878. PMID 31241843
- [Background] Kwok CS, Holland R, Gibbs S. Efficacy of topical treatments for cutaneous warts: a meta-analysis and pooled analysis of randomized controlled trials. Br J Dermatol. 2011 Aug;165(2):233-46. doi: 10.1111/j.1365-2133.2011.10218.x. Epub 2011 May 26. PMID 21219294